CLINICAL TRIAL: NCT06225557
Title: Comparison of Outcome Between the Implementation of Enhanced Recovery After Elective Cesarean Section Protocol (ERACS) Versus Traditional Methods
Brief Title: Comparison of Outcome Between (ERACS) Versus Traditional Methods in Elective CS
Acronym: ERACS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Marwa Abdelrehim Attia Mohamed, Assistant lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 383/08/2022
Record Dates: First submitted 2024-01-02; First posted 2024-01-26 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: ERAS

STUDY DESIGN:
Intervention Model Description: follow ERAS society guidelines recommendations in elective CESAREAN SECTION
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ERAS society guidlines (Experimental): The ERAS society guidelines for elective cesarean section will be followed.
  Interventions: Other: ERAS community recommendation
- Traditional methods (Experimental): Traditional methods in postoperative care for elective cesarean section will be followed.
  Interventions: Other: Traditional postoperative care

INTERVENTIONS:
Other: ERAS community recommendation — Enhanced recovery techniques including opioid sparing anesthesia in elective cesarean section
  Arms: ERAS society guidlines
Other: Traditional postoperative care — Usual anesthesia and analgesia in elective cesarean section.
  Arms: Traditional methods

SUMMARY:
The study is designed to evaluate the effect of implementing enhanced recovery after surgery (ERAS) protocol during elective cesarean section on patient's outcome measures.

DETAILED DESCRIPTION:
The study is designed to evaluate the effect of implementing enhanced recovery after surgery (ERAS) protocol during elective cesarean section on patient outcome measures. The primary outcome is the evaluation of inpatient postpartum recovery using the Obstetric Quality of Recovery 11 score (ObsQoR-11) at the time of discharge.

Secondary outcomes are the evaluation of peak numeric postoperative pain rating score within the postoperative hospital stay, total amount of postoperative opioid consumption, postoperative nausea, and vomiting impact score after 6 hours postoperatively and at time of discharge, patient satisfaction using Leiden perioperative care patient satisfaction questionnaire (LPPSq) at time of discharge, presence of post-cesarean ileus and Hospital length to achieve criteria for discharge.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ASA I to ASA II aged from 18 up to 40 years. With non-complicated pregnancy undergoing elective CS.

Exclusion Criteria:

* -Age less than 18 years
* Complications (wound infection, re-exploration, caesarean hysterectomies)
* Recent documented use of opioids Allergy to any drug used during the study.-
* Patients with severe heart diseases, cardiac arrhythmia and myocardial injury.
* uncontrolled diabetic patient
* Severe liver and kidney diseases
* Coagulation defect

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 106 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Obstetric Quality of Recovery 11 score (ObsQoR-11) | before discharge or during 24 hour postoperatively
  it is consisted of 11 questions covers four domains of recovery outcomes: physical comfort, emotional state, physical independence and care of the neonate, and pain ,each question taking score from 0 to 10 with 0 is the minimum score and 10 is the highest score and the maximum total score is 110 and the minimum total is 0 which is the worest quality of recovery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad EZ Mahran, professor, Principal Investigator — Faculty of Medicine, Minia University